CLINICAL TRIAL: NCT00288119
Title: Genetic and Environmental Determinants of Barrett's Esophagus and Esophageal Adenocarcinoma
Brief Title: Genetic Determinants of Barrett's Esophagus and Esophageal Adenocarcinoma
Acronym: FBE
Status: Recruiting | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Washington University School of Medicine (Other); Fred Hutchinson Cancer Center (Other); University of Washington (Other); Mercy Medical Center (Other); Johns Hopkins University (Other); Mayo Clinic (Other); University of North Carolina, Chapel Hill (Other); The Cleveland Clinic (Other); University of Pennsylvania (Other); Columbia University (Other); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: R01DK070863 (NIH); NIH IK24DK02800; NCT00058877 (obsolete NCT alias)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Barrett's Esophagus; Esophageal Neoplasm
Keywords: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Samples from + families with 3 or members diagnosed with BE or ECA will be sent to our NIH approved Biorepository and this repository is designed to help all researchers performing studies on the genetic basis of diseases.
  Biospecimens, brushings and biopsies, will be obtained via snap frozen at bedside and stored for future research assays at Case Western Reserve Biorepository.
  Balloon Capsule Device Tips are sent to the University Hospitals Transnational Laboratory in Cleveland. The tips are processed for process of assay of DNA and RNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Cases: Patients with Barrett's esophagus undergoing surveillance or patients with esophageal adenocarcinoma and esophagogastric junctional adenocarcinoma undergoing EGD
  Interventions: Device: Balloon Capsule Device; Procedure: Endoscopy
- EGD Screening: Patients scheduled for clinically indicated EGD for GERD who meet ACG criteria for BE screening
  Interventions: Device: Balloon Capsule Device; Procedure: Endoscopy
- Colon Screening: Patients scheduled for screening colonoscopy who have not had EGD and meet clinically indicated criteria for BE screening
  Interventions: Device: Balloon Capsule Device; Procedure: Endoscopy
- Controls: Patients scheduled for EGD who do not meet criteria for screening
  Interventions: Device: Balloon Capsule Device; Procedure: Endoscopy

INTERVENTIONS:
Device: Balloon Capsule Device — The Esophageal Sampling Device BESD-001 is a non-endoscopic balloon capsule catheter for obtaining an esophageal mucosal sample. At the distal end of the catheter there is a silicone capsule textured balloon assembly. The textured balloon is initially inverted with vacuum for patient to swallow the capsule but then is inflated with 5.6 cc of air (5 cc syringe withdrawn maximally) to a 16-18 mm diameter in order to contact the lumen of the esophagus to collect a sample. The balloon has a textured surface, which enhances the collection of the esophageal sample. Following sample collection the textured balloon is inverted back into the hollow capsule component via syringe draw vacuum in order to maximize & protect the site-specific sample collection.
  Other Names: Esophageal Sampling Device BESD-001
Procedure: Endoscopy — An upper endoscopy is a procedure used to visually examine your upper digestive system with a tiny camera on the end of a long, flexible tube.
  Other Names: EGD

SUMMARY:
The overall objectives of this BETRNet Research Center (RC) are:

1. to conduct a rigorous, integrated spectrum of transdisciplinary human research in Barrett's esophagus (BE) and esophageal adenocarcinoma (ECA)
2. to increase the biological understanding of key observations made by our clinical researchers;
3. to translate knowledge derived from genetic, epigenetic, and transcriptome research to solving clinical dilemmas in detection, prognosis, prevention, and therapy of BE in order to prevent EAC and improve the outcomes of EAC;
4. to foster a transdisciplinary and translation research culture and to effectively expand and enhance scientific research focused on BE and EAC;
5. to evaluate research and transdisciplinary programs and to continuously improve research, productivity and enhance translational implementation. These objectives build and synergize on existing multi-institutional collaborative networks and the considerable clinical, basic science, and translational expertise available at our institutions, focusing on improving the outcomes of patients with BE and EAC. The overarching organization framework for this RC proposal is 1) to focus laboratory research on understanding the genetic susceptibility, genomic and epigenetic changes that influence the development of BE and EAC; and 2) to then translate laboratorydiscoveries into clinical applications for effective detection, molecular risk stratification, and prevention of progression from BE to EAC.

DETAILED DESCRIPTION:
This research will eventually lead to the identification of inherited genetic changes that cause Barrett's esophagus and esophageal cancer. It will help the investigators develop better methods for preventing or identifying esophageal cancer at an early curable stage.

The capsule can be swallowed with a few sips water. Once the capsule is advanced to 45-50 cm from the incisors and reaches the stomach the balloon is inflated to a size of 16 mm with 5.5 cc air. It is withdrawn until a tug is felt to locate the gastroesophageal junction (GEJ). The inflated balloon is then pulled back 3 to 5 cm to sample the distal esophagus, then completely deflated to cause inversion of the biospecimen into its protective capsule, and then withdrawn. The balloon is re-inflated outside the patient and the obtained sample is clipped with scissors into a vial and frozen. The collected biospecimen will be stored frozen for later DNA extraction and assay. The vials will be labeled with a coded sample number. In a pilot study of 120 subjects this capsule esophageal sampling was performed with no adverse events reported. Similar esophageal sampling devices have been reported on over 1600 patients with no adverse events.

All patients will also undergo standard EGD. Patients with BE or EAC will have standard of care surveillance and diagnostic biopsies. All cases and controls will have research esophageal brushings from the BE/EAC and distal esophagus/gastric cardia, respectively. Cases and controls will also obtain research brushings from the proximal normal squamous esophagus. Research mucosal biopsies will also be obtained from the BE and EAC epithelium as well as normal stomach and duodenum in cases and from the gastric cardia and the distal squamous esophagus as well as normal stomach and duodenum in controls. Biopsies from BE and EAC will be directed by using high definition narrow band imaging. Biospecimens, brushings and biopsies, will be snap frozen at bedside and stored for future research assays. Although we do not anticipate any problems with our non-endoscopic balloon screening, these archived pathology samples and snap frozen samples will be available for assay in case we fail to detect our markers in patients with BE diagnosed at EGD or experience a high false positive rate. Subjects who undergo non-endoscopic sampling of the distal esophagus will be asked questions that rate their discomfort on a Likert scale and also asked questions comparing the non-endoscopic sampling study with an EGD.

ELIGIBILITY:
Eligible cases will be defined as those patients and their family members who meet the following criteria:

* Barrett's esophagus confirmed by review of pathology and endoscopy report or adenocarcinoma of the esophagus or family members of person with Barrett's esophagus or adenocarcinoma of the esophagus.
* Male or female age 18 or older at time of enrollment or male or female less than 18 years of age at time of enrollment with parental consent.
* Ability to give informed consent, if patient is age 18 or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Barrett's esophagus or adenocarcenoma of the esophagus whose medical care is at the participating institutions, are referred from outside institutions, or who contact the participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-10-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Assay of DNA and RNA markers | 1 week
  The Balloon tip is collected and sent to the PacificDx Laboratory in Irvine California to test for DNA extraction

SECONDARY OUTCOMES:
Score of tolerability and acceptability | 1 minute after procedure
  6 item scale rating scale using scale of 1-10 where 1 is no worries to 10 being severe to rate Tolerability; and a 3 item scale rating the acceptability of Balloon Capsule Device using strongly agree to strongly disagree rating

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Chak, MD, Principal Investigator — University Hospitals Cleveland Medical Center, CWRU, Cleveland, OH; Gary W Falk, MD, MS, Principal Investigator — University of Pennsylvania; William Grady, MD, Principal Investigator — Fred Hutchinson Cancer Research Center, UWMC, Seattle, WA; Nicholas J Shaheen, M.D., Principal Investigator — University of North Carolina, Chapel Hill; Ganapathy Prasad, M.D., Principal Investigator — Mayo Clinic; Marcia Canto, M.D., Principal Investigator — Johns Hopkins University; John Dumont, D.O., Principal Investigator — University Hospitals Cleveland Medical Center; Prashanthi Thota, M.D., Principal Investigator — The Cleveland Clinic; Jean Wang, MD, Principal Investigator — Washington University School of Medicine; Julian Abrams, MD, Principal Investigator — Columbia University; Andrew Kaz, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (10):
- United States (10):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, UWMC, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Douville C, Moinova HR, Thota PN, Shaheen NJ, Iyer PG, Canto MI, Wang JS, Dumot JA, Faulx A, Kinzler KW, Papadopoulos N, Vogelstein B, Markowitz SD, Bettegowda C, Willis JE, Chak A. Massively Parallel Sequencing of Esophageal Brushings Enables an Aneuploidy-Based Classification of Patients With Barrett's Esophagus. Gastroenterology. 2021 May;160(6):2043-2054.e2. doi: 10.1053/j.gastro.2021.01.209. Epub 2021 Jan 22. PMID 33493502
- [Derived] Moinova HR, Verma S, Dumot J, Faulx A, Iyer PG, Canto MI, Wang JS, Shaheen NJ, Thota PN, Aklog L, Willis JE, Markowitz SD, Chak A. Multicenter, Prospective Trial of Nonendoscopic Biomarker-Driven Detection of Barrett's Esophagus and Esophageal Adenocarcinoma. Am J Gastroenterol. 2024 Nov 1;119(11):2206-2214. doi: 10.14309/ajg.0000000000002850. Epub 2024 Apr 30. PMID 38686933
- [Derived] Chak A, Chen Y, Vengoechea J, Canto MI, Elston R, Falk GW, Grady WM, Guda K, Kinnard M, Markowitz S, Mittal S, Prasad G, Shaheen N, Willis JE, Barnholtz-Sloan JS. Variation in age at cancer diagnosis in familial versus nonfamilial Barrett's esophagus. Cancer Epidemiol Biomarkers Prev. 2012 Feb;21(2):376-83. doi: 10.1158/1055-9965.EPI-11-0927. Epub 2011 Dec 16. PMID 22178570